CLINICAL TRIAL: NCT00683111
Title: Famotidine Compared With Esomeprazole in the Prevention of Ulcer Complications in Patients With Acute Coronary Syndrome or Myocardial Infarction
Brief Title: Prevention of Gastrointestinal Bleeding in Patients With Severe Ischemic Heart Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ruttonjee Hospital (Other)
Responsible Party: Principal Investigator, Fook-Hong Ng, SMO, Ruttonjee Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HKEC-2007-176
Record Dates: First submitted 2008-05-21; First posted 2008-05-23 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2012-06

CONDITIONS: Acute Coronary Syndrome; Acute Myocardial Infarction
Keywords: acute coronary syndrome; acute myocardial infarction; aspirin; clopidogrel; heparin; thrombolytic; famotidine; esomeprazole
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Esomeprazole; Famotidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): oral esomeprazole 20 mg daily
  Interventions: Drug: esomeprazole 20 mg daily
- 2 (Active Comparator): oral famotidine 40mg daily
  Interventions: Drug: famotidine 40 mg daily

INTERVENTIONS:
Drug: esomeprazole 20 mg daily — oral famotidine 40 mg daily vs. oral esomeprazole 20 mg daily for up to 12 months
  Arms: 1
Drug: famotidine 40 mg daily — oral famotidine 40 mg daily vs. oral esomeprazole 20 mg daily for up to 12 months
  Arms: 2

SUMMARY:
Aspirin and clopidogrel +/- heparin or thrombolytic co-therapy is well established and effective treatment for unstable cardiac patients. However, the major complication was gastrointestinal bleeding (GIB) due to peptic ulcer. In the prevention of GIB, anti-ulcer drug either H2-receptor antagonist (H2RA) and proton pump inhibitor (PPI) were commonly prescribed. There has been no prospective controlled study to compare the efficacy of these two classes of anti-ulcer drugs.

ELIGIBILITY:
Inclusion Criteria:

* patients admitted for acute coronary syndrome or acute myocardial infarction requiring active treatment with aspirin clopidogrel and (enoxaparin or thrombolytics.)

Exclusion Criteria:

* known active peptic ulcer disease or gastrointestinal within 8 wk
* known iron deficiency anemia with Hb < 10 gm/dl
* mechanical ventilation
* active cancer, liver cirrhosis, end-stage renal failure
* life expectancy < 1 yr
* known allergic to aspirin, clopidogrel, enoxaparin famotidine or esomeprazole
* pregnancy, lactation, child-bearing potential in the absence of contraception,
* co-prescription of NSAID, corticosteroid, or warfarin
* non-oral feeding or impaired GI absorption e.g. vomiting
* already on proton pump inhibitor for > 1 day or another clinical trial drug for ulcer disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2008-07; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
ulcer complication (bleeding/perforation/obstruction) | up to 12 months

SECONDARY OUTCOMES:
Termination of anti-ischemic drug due to ulcer complications; TIMI severity of GI bleeding; Major adverse cardiac event (composite of death from CV causes, recurrent nonfatal MI, or stroke); | up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Fook Hong Ng, MBBS, Principal Investigator — Ruttonjee Hospital
Locations (1):
- Ruttonjee Hospital, Hong Kong, China

REFERENCES:
- [Derived] Ng FH, Tunggal P, Chu WM, Lam KF, Li A, Chan K, Lau YK, Kng C, Keung KK, Kwan A, Wong BC. Esomeprazole compared with famotidine in the prevention of upper gastrointestinal bleeding in patients with acute coronary syndrome or myocardial infarction. Am J Gastroenterol. 2012 Mar;107(3):389-96. doi: 10.1038/ajg.2011.385. Epub 2011 Nov 22. PMID 22108447